CLINICAL TRIAL: NCT05555615
Title: A 52-Week Open-Label Extension Study of Pimavanserin in Children and Adolescents With Irritability Associated With Autism Spectrum Disorder (ASD)
Brief Title: Extension Study of Pimavanserin in Irritability Associated With Autism Spectrum Disorder
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study was terminated for business reasons and not due to safety concerns.
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACP-103-070
Record Dates: First submitted 2022-08-30; First posted 2022-09-27 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Irritability Associated With Autism Spectrum Disorder
MeSH Terms: interventions — pimavanserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pimavanserin (Experimental): Pimavanserin once daily. All patients will receive the pimavanserin low dose (patients aged 5 to 12 years: 10 mg/day pimavanserin; patients aged 13 to 17 years: 20 mg/day) the first 2 weeks of the study. Thereafter, the dose may be increased to the high dose (5 to 12 years: 20 mg/day; 13 to 17 years: 34 mg/day) based on the Investigator's assessment of clinical response.
  After Week 2 and up to Week 20, dose adjustments are allowed at any clinic visit based on the Investigator's assessment of clinical response and tolerability. No further dose adjustments are allowed after Week 20.
  Interventions: Drug: Pimavanserin

INTERVENTIONS:
Drug: Pimavanserin — Pimavanserin given once daily, as capsule of 10, 20, or 34 mg dose strength, respectively, according to the patient's age
  Other Names: Nuplazid

SUMMARY:
52-week, open-label extension study of double-blind study ACP-103-069 to determine the long-term safety and tolerability of pimavanserin for the treatment of irritability associated with ASD in children and adolescents (aged 5 to 17 years).

ACP-103-069 is a 6-week, randomized, double-blind, fixed-dose, placebo controlled, parallel group study of pimavanserin in children and adolescents with irritability associated with autism spectrum disorder (ASD).

DETAILED DESCRIPTION:
This study will be conducted as a 52-week, open-label extension study of the antecedent double-blind study to determine the long-term safety and tolerability of pimavanserin for the treatment of irritability associated with ASD in children and adolescents (5 through 17 years old at the time of enrolling into the antecedent double-blind study).

ELIGIBILITY:
INCLUSION CRITERIA:

* Has completed the treatment period of study ACP-103-069
* Informed consent prior to the conduct of any study procedures
* Continues to be both clinically stable and not at imminent risk of suicide or injury to self, others, or property
* Continues to be medically stable at enrollment
* For female patients only: unable to become pregnant or agree to use a highly effective non-hormonal method of contraception. Females of childbearing potential must have a negative pregnancy test

EXCLUSION CRITERIA:

* Patient or parent/legally accepted representative is judged by the Investigator to be inappropriate for the study
* Requires treatment with a medication prohibited by the protocol, including concomitant psychotropic drugs targeting irritability, including those used off-label (clonidine, guanfacine, and propranolol; lithium, valproate), medications that prolong the QT interval; and strong cytochrome P450 (CYP) 3A4 enzyme (CYP3A4) inhibitors and inducers
* At a significant risk of suicide, or is a danger to self or others
* At risk of significant violent behavior to the extent that participation would pose an undue risk to other patients, caregivers, or others
* Positive urine drug test
* Serious and/or unstable psychiatric, neurologic, cardiovascular, respiratory, gastrointestinal, renal, hepatic, hematologic, or other medical disorder, including cancer or malignancies
* Any change in medical or treatment status that may increase the risk associated with taking pimavanserin, would interfere with safety assessments, or would confound the interpretation of study results
* Clinically significant abnormal ECG of protocol-defined cardiac conduction abnormalities
* Weight <15 kg
* Additional inclusion/exclusion criteria apply. Subjects will be evaluated at screening to ensure that all criteria for study participation are met.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 209 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (18):
  - Southwest Autism Research and Resource Center, Phoenix, Arizona
  - Cortica Inc. (Glendale), Glendale, California
  - Cortica Inc., San Rafael, California
  - 1st Allergy and Clinical Research Group, d/b/a IMUNOe Research Centers, Centennial, Colorado
  - Children's Research Institute, Washington D.C., District of Columbia
  - The EHS Medical Practice, PA, D/B/A Sarkis Clinical Trials, Gainesville, Florida
  - APG Research, LLC, Orlando, Florida
  - AMR Baber Research Incorporated, Naperville, Illinois
  - Clinical Research of Southern Nevada, LLC, Las Vegas, Nevada
  - ERG Clinical Research - New York, PLLC DBA Richmond Behavioral Associates, Staten Island, New York
  - Quest Therapeutics of Avon Lake dba Haidar Almhana Nieding LLC, Avon Lake, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Relaro Medical Trials, LLC, Dallas, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - AIM Trials, LLC, Plano, Texas
  - Eastside Therapeutic Resource, Inc. dba Core Clinical Research, Everett, Washington
- Australia (3):
  - Children's Health Queensland Hospital and Health Service, South Brisbane, Queensland
  - Monash Health, Clayton, Victoria
  - Murdoch Children's Research Institute, Parkville, Victoria
- France (4):
  - Centre Hospitalier Charles Perrens, Bordeaux
  - Centre de Ressources Autisme Rhône-Alpes - Center Hospitalier le Vinatier, Bron
  - CHU de Nantes, Nantes
  - L'Assistance Publique - Hôpitaux de Paris, labélisé Institut Carnot, Paris
- Hungary (3):
  - Magyarországi Református Egyház Bethesda Gyermekkórháza, Budapest
  - Békés Megyei Központi Kórház, Gyula
  - Szegedi Tudományegyetem, Szeged
- Italy (6):
  - La Nostra Famiglia - Scientifica IRCCS Eugenio Medea, Bosisio Parini, LC
  - Policlinico Riuniti - Azienda Ospedaliero Universitaria, Foggia
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Fondazione Istituto Neurologico Nazionale Casimiro Mondino - IRCCS, Pavia
  - Fondazione PTV - Policlinico Tor Vergata, Rome
  - Azienda Ospedaliera Universitaria Integrata di Verona (AOUI), Verona
- Poland (6):
  - Gdańskie Centrum Zdrowia Sp. z o.o., Gdansk
  - Centrum Badań Klinicznych PI-House Sp. z o.o., Gdansk
  - NAVICULA - Centrum Diagnozy i Terapii Autyzmu, Lodz
  - Ginemedica Sp. Zoo, S. K., Wroclaw
  - Centrum Neuropsychiatrii Neuromed SP ZOZ, Wroclaw
  - MedicMental Indywidualna Specjalistyczna Praktyka Lekarska Monika Szewczuk-Boguslawska, Wroclaw
- Serbia (4):
  - Institute of Mental Health, Belgrade
  - University Clinical Center Kragujevac, Clinic for Psychiatry, Kragujevac
  - University Clinical Center Nis, Center for Mental Health, Niš
  - Clinical Center of Vojvodina, Clinic for Psychiatry, Novi Sad
- Spain (4):
  - Hospital General de Alicante, Alicante
  - Institut Global d´Atenció Integral del Neurodesenvolupament (IGAIN), Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label extension study of the antecedent double-blind study ACP-103-069. Patients were eligible for this study if they had completed the treatment period of study ACP-103-069.
Groups:
- Pimavanserin: Pimavanserin once daily administered using age-based dosing:
  * pimavanserin low dose during Weeks 1 and 2 (age 5 to 12 years: 10 mg/day; age 13 to 17 years: 20 mg/day)
  * pimavanserin high dose from Week 3 onwards (5 to 12 years: 20 mg/day; 13 to 17 years: 34 mg/day) based on the investigator's assessment of clinical response Dose adjustments were allowed after Week 2 and up to Week 20, based on the investigator's assessment of clinical response and tolerability.
Period: Overall Study
Arm/Group | Pimavanserin
Started | 209
Completed | 67
Not Completed | 142
Not completed — Adverse Event | 7
Not completed — Lack of Efficacy | 12
Not completed — Lost to Follow-up | 10
Not completed — Noncompliance with study drug | 5
Not completed — Physician Decision | 2
Not completed — Study terminated by sponsor | 80
Not completed — Prohibited medication use | 2
Not completed — Withdrawal by Subject | 20
Not completed — Not further specified | 4

BASELINE CHARACTERISTICS:
Population: All patients enrolled and treated
Arm/Group | Pimavanserin
Number analyzed (Participants) | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.1 (3.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 163
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 24
  White | 158
  More than one race | 0
  Unknown or Not Reported | 16
Region of Enrollment [Number; unit: participants]
  Hungary | 17
  United States | 98
  Poland | 55
  Italy | 9
  France | 11
  Serbia | 9
  Australia | 6
  Spain | 4

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events
Description: Number (%) of patients with treatment emergent adverse events
Time Frame: 52 weeks
Population: All patients enrolled and treated
Measure: Count of Participants; unit: Participants
Groups:
- Pimavanserin: Pimavanserin once daily. All patients will receive the pimavanserin low dose (patients aged 5 to 12 years: 10 mg/day pimavanserin; patients aged 13 to 17 years: 20 mg/day) the first 2 weeks of the study. Thereafter, the dose may be increased to the high dose (5 to 12 years: 20 mg/day; 13 to 17 years: 34 mg/day) based on the Investigator's assessment of clinical response.
  After Week 2 and up to Week 20, dose adjustments are allowed at any clinic visit based on the Investigator's assessment of clinical response and tolerability. No further dose adjustments are allowed after Week 20.
  Pimavanserin: Pimavanserin given once daily, as capsule of 10, 20, or 34 mg dose strength, respectively, according to the patient's age
Arm/Group | Pimavanserin
Number analyzed (Participants) | 209
Participants | 132

2. Secondary Outcome: Aberrant Behavior Checklist-Irritability (ABC-I) and Clinical Global Impression-Improvement (CGI-I) Response Rate
Description: The response rate was defined as the proportion of patients with at least 25% reduction from baseline to Week 52 in ABC-I and a CGI-I of irritability score of 1 (very much improved) or 2 (much improved) at Week 52, compared to baseline.
  Baseline was the baseline of the antecedent double-blind study APC-103-069. The ABC is a parent/caregiver-rated scale comprised of 5 subscales encompassing 58 items. Subscales are irritability, lethargy, stereotypic behavior, hyperactivity, and inappropriate speech. Items are rated on a 4-point Likert scale ranging from 0 (not at all a problem) to 3 (the problem is severe), with higher scores indicating more severe problems. Subscale scores are calculated by summing the items within that subscale.
  The CGI-I is a clinician-rated, 7-point scale to assess how much the patient's illness (here: the patient's irritability) has changed relative to baseline. Scores range from 1 (very much improved) to 7 (very much worse).
Time Frame: 52 weeks
Population: All patients enrolled and treated
Measure: Count of Participants; unit: Participants
Arm/Group | Pimavanserin
Number analyzed (Participants) | 209
Participants | 51

ADVERSE EVENTS:
Time Frame: 52 weeks (study terminated early by the sponsor)
Arm/Group | Pimavanserin
All-Cause Mortality (participants affected / at risk) | 0/209
Serious Adverse Events (participants affected / at risk) | 5/209
Other Adverse Events (participants affected / at risk) | 66/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin (N=209)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1)
Heart rate irregular (Investigations) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin (N=209)
Vomiting (Gastrointestinal disorders) | 15 (17)
Pyrexia (General disorders) | 11 (12)
Upper respiratory tract infection (Infections and infestations) | 21 (29)
Nasopharyngitis (Infections and infestations) | 13 (19)
Headache (Nervous system disorders) | 14 (16)

LIMITATIONS AND CAVEATS:
The study was terminated early by the Sponsor due to lack of efficacy in the antecedent double-blind study (ACP-103-069).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to their own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the Sponsor for review and comment. The sponsor has 60 days to review and comment.

DOCUMENTS (2):
  • Study Protocol (2024-02-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT05555615/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-19): https://cdn.clinicaltrials.gov/large-docs/15/NCT05555615/SAP_001.pdf